CLINICAL TRIAL: NCT03932968
Title: Observational Study of Epigastric Symptoms Chronicles, the Rise of the Line of Clips and Their Management in Obese Patients One Year Later Sleeve Gastrectomy
Brief Title: Clip Ascent and Sleeve Gastrectomy
Acronym: POST-SLEEVE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI17015J; 2017-A01608-45 (Other: ANSM)
Record Dates: First submitted 2018-01-02; First posted 2019-05-01 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Sleeve Gastrectomy; Obesity
Keywords: sleeve gastrectomy; clip ascent; oesogastric reflux; sleeve gastrectomy follow-up
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic pain: For patients with gastric symptoms such as retrosternal burning, regurgitations, and epigastric pain, a pH-metry during 24 hours will be performed.
  Interventions: Procedure: pH-metry during 24 hours
- Control: patients after a sleeve gastrectomy without symptomatic pain

INTERVENTIONS:
Procedure: pH-metry during 24 hours — For patients with gastric symptoms such as retrosternal burning, regurgitations, and epigastric pain, a pH-metry will be performed
  Groups: Symptomatic pain

SUMMARY:
This is a single institution study. All patients, one year after sleeve gastrectomy will be included. All will have a CT scan looking for clip ascent. For patients with chronic gastric symptoms such as retrosternal burning, regurgitations, and epigastric pain, a pH-metry will be performed. Those symptoms appeared at least 6 months after the surgery. A second consultation is done one year after. The aim of the study is to correlate clip ascent, pyrosis proved by ph-metry and epigastric symptoms after sleeve gastrectomy. The demographic data collection confirms the definition of clip ascent, define its frequency, and look for correlation with the median weight loss.

DETAILED DESCRIPTION:
There is a strong association between gastric reflux and obesity. A severe reflux is a contraindication for a sleeve gastrectomy for some surgeons. However the impact of sleeve gastrectomy on reflux is not clear. A de novo reflux is described for 2 to 18% of patients and many patients have unclear epigastric symptoms. One of the cause could be clip ascent which could justify a second surgery. This is a single institution study. All patients, one year after sleeve gastrectomy will be included. All will have a CT scan looking for clip ascent. For patients with gastric symptoms such as retrosternal burning, regurgitations, and epigastric pain, a pH-metry will be performed. A second consultation is done one year after. The aim of the study is to correlate clip ascent, pyrosis proved by ph-metry and epigastric symptoms after sleeve gastrectomy. The demographic data collection, confirms the definition of clip ascent, define its frequency, and look for correlation with the median weight loss. A medical information note is given to every patient at the first consultation.

ELIGIBILITY:
Inclusion Criteria:

* sleeve gastrectomy operated for at least 1 year

Exclusion Criteria:

* acute abdominal pain,
* epigastric pain occuring after the surgery (no 6 months delay),
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients operated on a sleeve gastrectomy realizing their consultation at 12 months post sleeve
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2017-12-17 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Measure of clip ascent | 12 months
  All patients at one year after a sleeve gastrectomy will be included. They will all have a CT scan and symptomatic patients will have a phmetry. Observational between epigastric symptoms, clip ascent at one year after a sleeve gastrectomy.

SECONDARY OUTCOMES:
Frequency of clip ascent | 18 months
  Clip ascent is noticed after sleeve surgery but data about it are unknown
Oesogastric reflux proved by phmetry | 12 months
  The frequency of oesogastric reflux proved by phmetry at 12 months after surgery is unknown

CONTACTS AND LOCATIONS:
Overall Officials: PASCALE KARILA-COHEN, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Bichat, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided